CLINICAL TRIAL: NCT01843205
Title: Buspirone as a Candidate Medication for Methamphetamine Abuse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Craig Rush, Professor, University of Kentucky
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: R21DA035481 (NIH); R21DA035481 (NIH)
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Methamphetamine Dependence; Methamphetamine Abuse
MeSH Terms: interventions — Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be maintained on placebo.
  Interventions: Drug: Methamphetamine; Drug: Placebo
- Buspirone (Experimental): Subjects will be maintained on buspirone.
  Interventions: Drug: Methamphetamine; Drug: Placebo

INTERVENTIONS:
Drug: Methamphetamine — The pharmacodynamic effects of methamphetamine will be determined during placebo and buspirone maintenance.
Drug: Placebo — The pharmacodynamic effects of placebo methamphetamine will be determined during placebo and buspirone maintenance.

SUMMARY:
Methamphetamine use disorders are an unrelenting public health concern. Intensive research efforts have yielded behavioral interventions that reduce methamphetamine use, however, these interventions are not universally effective and treatment effects diminish over time. Development of a pharmacotherapy that enhances the efficacy of these interventions is a priority for the National Institute on Drug Abuse. This study proposes to determine the impact of buspirone maintenance on self-administration of methamphetamine. These preliminary data will be used to support further research developing buspirone as a pharmacotherapy for methamphetamine use disorders. The investigators hypothesize that buspirone will attenuate the reinforcing effects of methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime methamphetamine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to methamphetamine or buspirone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Buspirone: Subjects were maintained on placebo for 7 days, then they were crossed over to 45 mg buspirone daily for 7 days.
- Buspirone Then Placebo: Subjects were maintained on 45 mg buspirone daily for 7 days, then they were crossed over to placebo for 7 days.
Period: First Treatment (11 Days)
Arm/Group | Placebo Then Buspirone | Buspirone Then Placebo
Started | 5 | 4
Completed | 4 (4 completing subjects switched to buspirone for Condition 2.) | 4 (4 completing subjects switched to placebo for Condition 2.)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Treatment (11 Days)
Arm/Group | Placebo Then Buspirone | Buspirone Then Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Completing Participants: All subjects who completed the study.
Arm/Group | Completing Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Methamphetamine Doses Self-Administered
Description: The reinforcing effects of methamphetamine will be determined during placebo and buspirone treatment using a modified progressive ratio procedure in which subjects are offered the opportunity to earn previously sampled doses of methamphetamine. Each ratio completed on the task will earn 1/10th of the sampled dose.
Time Frame: One test per methamphetamine dose level per intervention for each participant over his/her approximate 25 day inpatient admission
Measure: Mean (Standard Error); unit: Number of Methamphetamine Doses
Groups:
- Placebo: Subjects were maintained on placebo for 7 days.
- Buspirone: Subjects were maintained on 45 mg buspirone daily for 7 days.
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
Number of Methamphetamine Doses
  Placebo Methamphetamine | 1.25 (1.25) | 0 (0)
  10 mg Methamphetamine | 6.13 (1.72) | 4 (1.78)
  30 mg Methamphetamine | 7.88 (1.42) | 7.5 (1.64)

2. Secondary Outcome: Peak Score on Sedative Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Sedative Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "sedative" items was summed to yield the Sedative Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both bupsirone and placebo conditions.
Time Frame: Subjects completed this measure at 15 minute intervals for 2 hours after sampling each methamphetamine dose under both buspirone and placebo maintenance conditions.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 3.38 (1.66) | 2.75 (1.42)
  10 mg Methamphetamine | 3.63 (1.08) | 3.75 (1.33)
  30 mg Methamphetamine | 3 (0.96) | 3.25 (1.10)

3. Secondary Outcome: Peak Score on Stimulant Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Stimulant Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "stimulant" items was summed to yield the Stimulant Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both bupsirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 5.63 (1.18) | 7.25 (2.14)
  10 mg Methamphetamine | 9.88 (1.59) | 9.25 (1.78)
  30 mg Methamphetamine | 11.38 (1.59) | 13 (2.14)

4. Secondary Outcome: Peak Ratings of "Active, Alert, Energetic" on the Visual Analog Scale
Description: Subjects rated their feelings of "Active, Alert, Energetic" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 2.13 (1.54) | 8.75 (8.75)
  10 mg Methamphetamine | 19 (9.51) | 14.5 (10.36)
  30 mg Methamphetamine | 35 (11.25) | 29.25 (10.30)

5. Secondary Outcome: Peak Ratings of "Any Effect" on the Visual Analog Scale
Description: Subjects rated their feelings of "Any Effect" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.75 (0.49) | 10 (9.12)
  10 mg Methamphetamine | 25.75 (8.25) | 21.5 (8.35)
  30 mg Methamphetamine | 34.38 (11.51) | 33 (10.04)

6. Secondary Outcome: Peak Ratings of "Bad Effects" on the Visual Analog Scale
Description: Subjects rated their feelings of "Bad Effects" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.13 (0.13) | 1.5 (1.5)
  10 mg Methamphetamine | 7 (6.45) | 7.63 (4.04)
  30 mg Methamphetamine | 3.13 (3.13) | 8.38 (4.00)

7. Secondary Outcome: Peak Ratings of "Euphoric" on the Visual Analog Scale
Description: Subjects rated their feelings of "Euphoric" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.63 (0.63) | 0 (0)
  10 mg Methamphetamine | 4.88 (2.41) | 3.88 (2.81)
  30 mg Methamphetamine | 7.63 (4.31) | 8.5 (4.78)

8. Secondary Outcome: Peak Ratings of "Good Effects" on the Visual Analog Scale
Description: Subjects rated their feelings of "Good Effects" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.88 (0.64) | 9.63 (9.34)
  10 mg Methamphetamine | 21 (9.01) | 17.38 (10.36)
  30 mg Methamphetamine | 30.63 (12.04) | 31.5 (10.82)

9. Secondary Outcome: Peak Ratings of "High" on the Visual Analog Scale
Description: Subjects rated their feelings of "High" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.63 (0.63) | 10.5 (9.66)
  10 mg Methamphetamine | 22.13 (8.71) | 16.5 (10.51)
  30 mg Methamphetamine | 28.63 (10.80) | 31 (11.28)

10. Secondary Outcome: Peak Ratings of "Irregular/Racing Heartbeat" on the Visual Analog Scale
Description: Subjects rated their feelings of "Irregular/Racing Heartbeat" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.75 (0.75) | 8.5 (8.5)
  10 mg Methamphetamine | 10.63 (10.34) | 10.75 (9.92)
  30 mg Methamphetamine | 14.38 (11.33) | 16.13 (11.54)

11. Secondary Outcome: Peak Ratings of "Like Drug" on the Visual Analog Scale
Description: Subjects rated their feelings of "Like Drug" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.63 (0.63) | 9.63 (9.48)
  10 mg Methamphetamine | 22.63 (8.87) | 18.50 (10.77)
  30 mg Methamphetamine | 32.75 (11.82) | 30.50 (11.16)

12. Secondary Outcome: Peak Ratings of "Nauseous" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nauseous" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0 (0) | 0 (0)
  10 mg Methamphetamine | 6.38 (5.14) | 2.38 (2.38)
  30 mg Methamphetamine | 3.50 (2.50) | 5 (3.81)

13. Secondary Outcome: Peak Ratings of "Nervous/Anxious" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nervous/Anxious" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.88 (0.88) | 0 (0)
  10 mg Methamphetamine | 2.38 (1.69) | 1 (0.63)
  30 mg Methamphetamine | 4 (1.84) | 3.75 (2.66)

14. Secondary Outcome: Peak Ratings of "Willing to Pay For" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Pay For" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 1.63 (1.49) | 9.38 (8.82)
  10 mg Methamphetamine | 19.88 (9.65) | 17.75 (10.18)
  30 mg Methamphetamine | 34.00 (11.78) | 31.63 (10.99)

15. Secondary Outcome: Peak Ratings of "Performance Impaired" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Impaired" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.25 (0.25) | 0 (0)
  10 mg Methamphetamine | 2.13 (1.54) | 0 (0)
  30 mg Methamphetamine | 0 (0) | 1.38 (1.12)

16. Secondary Outcome: Peak Ratings of "Performance Improved" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Improved" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0 (0) | 9.25 (9.11)
  10 mg Methamphetamine | 15 (9.32) | 13.38 (10.60)
  30 mg Methamphetamine | 19.13 (12.24) | 22.75 (12.07)

17. Secondary Outcome: Peak Ratings of "Restless" on the Visual Analog Scale
Description: Subjects rated their feelings of "Restless" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 5 (5) | 0 (0)
  10 mg Methamphetamine | 3.13 (1.67) | 0.50 (0.50)
  30 mg Methamphetamine | 0.25 (0.25) | 1.13 (0.58)

18. Secondary Outcome: Peak Ratings of "Rush" on the Visual Analog Scale
Description: Subjects rated their feelings of "Rush" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.13 (0.13) | 10.25 (9.97)
  10 mg Methamphetamine | 21.63 (8.28) | 16.50 (10.57)
  30 mg Methamphetamine | 21.75 (11.04) | 26.13 (11.14)

19. Secondary Outcome: Peak Ratings of "Shaky/Jittery" on the Visual Analog Scale
Description: Subjects rated their feelings of "Shaky/Jittery" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0.13 (0.13) | 8.38 (7.69)
  10 mg Methamphetamine | 1.88 (1.32) | 0.75 (0.53)
  30 mg Methamphetamine | 2.88 (1.90) | 5.50 (2.33)

20. Secondary Outcome: Peak Ratings of "Sluggish/Fatigued/Lazy" on the Visual Analog Scale
Description: Subjects rated their feelings of "Sluggish/Fatigued/Lazy" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 1.5 (1.5) | 0 (0)
  10 mg Methamphetamine | 1.88 (1.49) | 2.88 (1.99)
  30 mg Methamphetamine | 3.13 (2.60) | 2.25 (2.25)

21. Secondary Outcome: Peak Ratings of "Stimulated" on the Visual Analog Scale
Description: Subjects rated their feelings of "Stimulated" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 1.25 (0.77) | 9.88 (9.31)
  10 mg Methamphetamine | 21.88 (8.86) | 17.88 (10.81)
  30 mg Methamphetamine | 21.50 (11.25) | 24.25 (11.23)

22. Secondary Outcome: Peak Ratings of "Willing to Take Again" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Take Again" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 1.25 (1.11) | 9.62 (9.34)
  10 mg Methamphetamine | 22.00 (9.03) | 20.63 (10.25)
  30 mg Methamphetamine | 35.00 (12.28) | 33.00 (10.62)

23. Secondary Outcome: Peak Ratings of "Talkative/Friendly" on the Visual Analog Scale
Description: Subjects rated their feelings of "Talkative/Friendly" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
units on a scale
  Placebo Methamphetamine | 0 (0) | 9.25 (8.69)
  10 mg Methamphetamine | 18.50 (10.10) | 13.75 (9.76)
  30 mg Methamphetamine | 26.00 (10.48) | 27.25 (10.24)

24. Secondary Outcome: Peak Diastolic Blood Pressure
Description: Diastolic blood pressure was measured with an automated monitor. Higher values represent greater diastolic pressure. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
mm Hg
  Placebo Methamphetamine | 77.50 (2.27) | 80.13 (3.93)
  10 mg Methamphetamine | 80.75 (2.52) | 83.00 (3.94)
  30 mg Methamphetamine | 83.80 (2.25) | 84.50 (2.95)

25. Secondary Outcome: Peak Systolic Blood Pressure
Description: Systolic blood pressure was measured with an automated monitor. Higher values represent greater systolic pressure. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
mm Hg
  Placebo Methamphetamine | 125.38 (3.84) | 125.00 (2.68)
  10 mg Methamphetamine | 131.25 (3.71) | 131.63 (3.72)
  30 mg Methamphetamine | 139.63 (4.18) | 137.13 (2.57)

26. Secondary Outcome: Peak Heart Rate
Description: Heart rate was measured with an automated monitor. Higher values represent greater heart rate. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
beats per minute
  Placebo Methamphetamine | 82.75 (6.65) | 81.25 (2.69)
  10 mg Methamphetamine | 86.13 (3.27) | 85.13 (5.00)
  30 mg Methamphetamine | 85.38 (5.90) | 90.63 (3.89)

27. Secondary Outcome: Peak Temperature
Description: Oral temperature was measured with an automated monitor. Higher values represent greater temperature. Peak scores were calculated from multiple assessments for each methamphetamine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: degrees Fahrenheit
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 8 | 8
degrees Fahrenheit
  Placebo Methamphetamine | 98.48 (0.07) | 98.41 (0.08)
  10 mg Methamphetamine | 98.44 (0.10) | 98.46 (0.05)
  30 mg Methamphetamine | 98.33 (0.07) | 98.43 (0.05)

ADVERSE EVENTS:
Time Frame: Approximately 25 days of inpatient admission
Groups:
- Placebo: All completing subjects who received placebo maintenance.
- Buspirone: All completing subjects who received buspirone maintenance.
Arm/Group | Placebo | Buspirone
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT01843205/Prot_SAP_000.pdf